CLINICAL TRIAL: NCT06194500
Title: An Open-label, Two-part Study of the Disposition and Absolute Bioavailability of [14C]-LY3549492 in Healthy Participants
Brief Title: A Study of Carbon-14-Labeled [14C]-LY3549492 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18348; J3H-MC-GZNC (Other: Eli Lilly and Company); U1111-1293-8652 (Other: UTN)
Record Dates: First submitted 2023-12-20; First posted 2024-01-08 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Healthy Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon-14-Labeled [14C]-LY3549492 - Part A (Experimental): Carbon-14-Labeled [14C]-LY3549492 administered as oral solution.
  Interventions: Drug: [14C]-LY3549492
- LY3549492 + [14C]-LY3549492 - Part B (Experimental): LY3549492 administered as oral solution followed 3 hours later by [14C] LY3549492 will be administered as intravenous (IV) infusion.
  Interventions: Drug: LY3549492; Drug: [14C]-LY3549492

INTERVENTIONS:
Drug: [14C]-LY3549492 — Administered as oral solution.
  Arms: Carbon-14-Labeled [14C]-LY3549492 - Part A
Drug: LY3549492 — Administered orally.
  Arms: LY3549492 + [14C]-LY3549492 - Part B
Drug: [14C]-LY3549492 — Administered as IV infusion.
  Arms: LY3549492 + [14C]-LY3549492 - Part B

SUMMARY:
The main purpose of this study is to measure how much of the study drug gets into the bloodstream and how long it takes the body to get rid of it. This study will be conducted in healthy males and has two parts. In Part A, participants will receive carbon-14 (14C) radiolabeled LY3549492 ([14C] LY3549492) given by mouth. In Part B, participants will receive LY3549492 by mouth. Three hours later, participants will receive [14C] LY3549492 given into a vein.

The radioactive substance C14 will be incorporated into the study drug to investigate the study drug and breakdown products to find out how much of these passes from blood into urine, stool, and breath.

The study will last about 2 months in Part A and about 1½ months in Part B. This includes screening, treatment, and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG).
* Participants who have safety laboratory test results within normal reference ranges, or results with acceptable deviations that are deemed not clinically significant by the investigator.
* Body mass index (BMI) within the range of 20.0 to 40.0 kilograms per meter squared (kg/m2), inclusive.
* Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Have known allergies to LY3549492, glucagon-like peptide-1 (GLP-1) non-peptide agonist (NPA)-related compounds or any components of the formulation as appropriate, or history of atopy.
* Have a clinical diagnosis of a long QT syndrome.
* Have any abnormality in the 12-lead ECG at screening that, in the opinion of the investigator, may increase the risk associated with participation in the study or may confound ECG data analysis.
* Have significant history of any current serious medical condition.
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis) or have an elevation in serum amylase or lipase (>1.0×Upper Limit Normal (ULN)).

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of Total Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose in Part A | Predose up to Day 24 postdose in Part A
  Urinary Excretion of Total Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose
Fecal Excretion of Total Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose in Part A | Predose up to Day 24 postdose in Part A
  Fecal Excretion of Total Radioactivity Over Time Expressed as a Percentage of the Total
Pharmacokinetic (PK): Area Under the Curve (AUC) for Oral Determination of Absolute Bioavailability (F) of LY3549492 in Part B | Predose up to Day 7 postdose in Part B
  PK: AUC for oral determination of absolute bioavailability (F) of LY3549492
PK: AUC for Intravenous (IV) Determination of Absolute Bioavailability (F) of LY3549492 in Part B | Predose up to Day 7 postdose in Part B
  PK: AUC for IV determination of absolute bioavailability (F) of LY3549492

SECONDARY OUTCOMES:
PK: Area Under the Concentration (AUC) for Radioactivity in Plasma and Whole Blood in Part A | Predose up to Day 24 postdose in Part A
  PK: AUC for radioactivity
PK: Maximum Concentration (Cmax) for Radioactivity in Plasma and Whole Blood in Part A | Predose up to Day 24 postdose in Part A
  PK: Cmax for radioactivity
PK: AUC of LY3549492 in Plasma in Part A | Predose up to Day 24 postdose in Part A
  PK: AUC of LY3549492 in plasma
PK: Cmax of LY3549492 in Plasma in Part A | Predose up to Day 24 postdose in Part A
  PK: Cmax of LY3549492 in plasma
Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable) in Part A | Predose up to Day 24 postdose in Part A
  Total radioactivity recovered in urine, feces, and expired air (if applicable) in Part A
Total Number of Metabolites and Identification of Metabolites of LY3549492 in Part A | Predose up to Day 24 postdose in Part A
  Total number of metabolites and identification of metabolites of LY3549492
PK: AUC of LY3549492, [14C]-LY3549492, and Total Radioactivity in Plasma in Part B | Predose up to Day 7 postdose in Part B
  AUC of LY3549492, [14C]-LY3549492, and total radioactivity in plasma in Part B
PK: Cmax of LY3549492, [14C]-LY3549492, and Total Radioactivity in Plasma in Part B | Predose up to Day 7 postdose in Part B
  Cmax of LY3549492, [14C]-LY3549492, and total radioactivity in plasma in Part B
Total Radioactivity Recovered in Urine and Feces in Part B | Predose up to Day 7 postdose in Part B
  Total radioactivity recovered in urine and feces in Part B

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 : Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Holbeck, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No